CLINICAL TRIAL: NCT04732702
Title: Effects of Contact Restrictions During the COVID-19 Pandemic on Newborns and Their Parents in Terms of Mother-infant Interaction, Parental Well-being, Expression and Methylation of Candidate Genes of Stress Signaling Pathways
Brief Title: Effects of Contact Restrictions During the COVID-19 Pandemic on Newborns and Their Parents
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, adjunct professor, medical doctor, University of Cologne
Other Study IDs: 20-1440
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Mother-Child Interaction
Keywords: stress response; neurodevelopment; newborn; SARS-CoV-2
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 buccal swabs with mucosal epithelial cells for RNA and DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There will be no intervention.

SUMMARY:
In the study, the researchers aim to investigate the impact of contact restrictions during the pandemic of coronavirus disease 2019 (COVID-19) caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) on newborns and their parents. At the onset of this COVID-19 pandemic, contact restrictions in Germany were introduced on March 16th, 2020. These included, among others, the ban on visits to hospitals. This also applied to visits by fathers of newborn children. In many hospitals, fathers were allowed to accompany the mother in the delivery room for birth, but had to leave the hospital before the mother was being transferred to the ward. Fathers were not allowed to visit their wives and newborns until discharge several days later.

The hypothesis of this study is that these contact restrictions have an influence on mother-infant interaction as well as on the psychological well-being of the parents. Furthermore, the investigators postulate that these restrictions additionally have a long-term effect on neonatal stress signaling pathways. For this purpose, children are studied, who were born during the period of strict contact restrictions from March, 16th to April, 30th, 2020. The children will be assessed at about six months of age.

DETAILED DESCRIPTION:
Due to the COVID-19 pandemic in spring 2020, the German government decided to impose strict contact restrictions to prevent an exponential increase in SARS-CoV-2-positive individuals. These included visiting regulations in hospitals from March 16th, 2020. These also applied to obstetrics departments in Cologne until April 30th, 2020. At the Obstetrics University Hospital Cologne as well as at the Protestant Hospital Cologne-Weyertal, fathers were allowed to be present in the delivery room for the birth of their newborns, but had to leave the hospital again before the mothers were being transferred to the obstetrics ward. The fathers could not see their newborn again until they were discharged a few days later. The consequences of these contact restrictions on the newborns and their parents have been little studied.

In a few hospitals, there were exceptions currently to the strict contact restrictions. These included the Hospital of the Augustinian Sisters in Cologne, where no visitation bans were imposed on fathers in the obstetrics department. With general precautions fathers were still allowed to accompany their newborns and mothers in the obstetric ward. The study of the newborns of this hospital enables the researchers to see whether the parents were nevertheless affected by the general changes in the living situation during a pandemic.

The phenomenon of "neonatal programming", which establishes the connection between formative influences in the neonatal period (e.g. pain or stress by separation of mothers) and disorders in later life (attention deficits, lack of concentration, learning difficulties) has received increasing attention in recent years. In particular, the search for molecular mechanisms that cause such programming has been the focus of scientific projects. In a delivery-room skin-to-skin study (deisy) conducted by this research group preterm infants were randomized to skin-to-skin contact or visual contact with their mothers. Significant differences were found in both mother-infant interaction at six months of age and the expression of candidate genes of stress signaling pathway.

An important regulatory mechanism for influencing the activity of certain genes in the long term is the methylation of their promoter region. This epigenetic regulatory mechanism plays an important role, so that the modulation of DNA methylation by events in the neonatal period could be responsible for a permanent determination of a certain infant phenotype. This methylation in candidate genes in the stress signaling pathway is currently investigated by the research team in healthy mature neonates born before the onset of the pandemic, and results are pending.

The aim of the present study is to investigate the impact of contact restrictions during the coronavirus pandemic on newborns and their parents.

Normally in healthy mother-infant-dyads without separation during the first postpartal hours, the mother has the best conditions to develop a high level of sensitivity. Sensitive maternal behavior favors the formation of optimal mother-infant interaction and is relevant for infant neurocognitive development. Due to the stressful situation caused by the separation of the father for several days, the psychological well-being of the parents as well as the optimal mother-child interaction could be negatively affected.

ELIGIBILITY:
Inclusion Criteria:

* birth from March, 16th, 2020 to April, 30th, 2020 with with subsequent stay for at least 48 hours in the obstetrics wards of the University Hospital of Cologne, the obstetrics department of the protestant hospital Köln-Weyertal or Hospital of Augustinian Sister's of Cologne
* mature newborn (38+0 to 41+6 weeks of gestational age)
* first child
* no separation of mother and child after birth
* informed consent
* good german language skills

Exclusion Criteria:

* multiples
* malformations or syndromes in the infant, reanimation after birth
* maternal psychological or severe physical illness

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consits of healthy mature newborns who were born during the time of strict contact restrictions from March, 16th to April, 30th, 2020. The recruitment will take place in three obstetric hospitals in Cologne (University Hospital of Cologne, Krankenhaus der Augustinnerinnen, evangelisches Krankenhaus Köln-Weyertal).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Analysis of the mother-child-interaction | at the age of six to nine months
  Mother-child interaction is investigated at the age of about six months using Mannheim Rating Scales. Therefore a five-minute-videotape of the mother changing the infant's diapers and playing with the infant is used. Mannheim Rating Scales is a good validated standardized observation instrument. Stimulation and response from the mother as well from the infant are being recorded. Different communication channels can be used by mother and child (vocal, facial or motor). All behaviors are analysed at intervals of five seconds (event coding). Then the values are formed from the sum of the coded events.The scale ranges from 0 to 60. If there is no interaction, the scale is 0. If there is an interaction in each interval (every 5 seconds in a 5 minute videotape), the scale is 60. The mother-child interaction is better if the scale is higher.

SECONDARY OUTCOMES:
Analysis of expression and methylation of candidate genes of stress signaling pathways from mucosal epithelial cells (buccal swab) | at the age of six to nine months
  RNA and DNA will be extracted from mucosal epithelial cells. The expression and methylation of candidate genes of the stress signaling pathways are investigated. The candidate genes are glucocorticoid receptor (NR3C1), corticotropin-releasing hormone receptor 1 (CRHR1) and 2 (CRHR2), serotonin receptors (1A and 2A), serotonin transporter (slc6a4) and vasopressin.
parental depression | at the infant's age of six to nine months
  Parental depression is assessed by the German long form of the Center for Epidemiological Studies Depression Scale (CES-D). It is a self-report questionnaire to measure depressive symptoms and it consists of 20 questions. For each question the response choice are assigned point values (how often a symptom occurred during the last week). The point values are summed to a total measure score. The score ranges from 0 to 60. Zero points represents no symptoms of depression, a score of 15 or higher is interpreted to indicate a risk of depression.
parental subjective distress caused by traumatic events | at the infant's age of six to nine months
  Parental subjective distress caused by traumatic events is assessed by the revised Impact of Event Scale (IES-R). It is a self-report questionnaire to measure subjective distress after a traumatic event and consists of 22 questions. Items are rated on a five point rating scale (from 0 to 4) and consists of three subscales (intrusion, hyperarousal and avoidance). The total score ranges from 0 to 88 and subscale scores can also be calculated. There is a cutoff score for the preliminary diagnosis of post-traumatic stress disorder, which is calculated by a formula (cutoff score, when X>0).
Social support | at the infant's age of six to nine months
  Social support is assessed with the short version of the F-SozU (Fragebogen zur sozialen Unterstützung,questionnaire on social support) scale (F-SozU K-22). The questionnaire records the subjectively perceived or anticipated support from the social environment. There are 22 items and the test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). The scale ranges from a minimum of 22 points to a maximum of 110 points. The higher the score, the better the subjectively perceived or anticipated support.
parental stress | at the infant's age of six to nine months
  Parental stress is assessed with the German form of the parenting stress index (PSI). It consists of 48 items. The test person can indicate the degree of agreement on a five-level Likert scale (from 1 = does not apply to 5 = applies completely). There are 12 subscales, each consisting of 4 items and the points on the Likert scale are added. In each subscale there can be a minimum of 4 and a maximum of 20 points. The higher the score,the higher the parental stress.
parental bonding | at the infant's age of six to nine months
  Parental Bonding is assessed with the parental bonding questionnaire (PBQ). It consists of 25 items and each itemis rated on a scale from 0 to 5 points (response range from "never" to "always"). There are four subscales and the point values of each subscale are summed to a total measure score. The four subscales are: impaired bonding,rejection and anger, anxiety about care, risk of abuse. The higher the score, the higher the risk of a disorder in each area of the subscale.
breastfeeding | at the infant's age of six to nine months
  The breastfeeding of the child is surveyed by a questionnaire according to World Health Organization criteria (early initiation of breastfeeding, exclusive breastfeeding for the first six months of life and introduction of complementar foods at 6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Cologne, Department of Neonatology, Cologne, Northrhine-westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehler K, Hucklenbruch-Rother E, Trautmann-Villalba P, Becker I, Roth B, Kribs A. Delivery room skin-to-skin contact for preterm infants-A randomized clinical trial. Acta Paediatr. 2020 Mar;109(3):518-526. doi: 10.1111/apa.14975. Epub 2019 Sep 16. PMID 31423649
- [Background] Hucklenbruch-Rother E, Vohlen C, Mehdiani N, Keller T, Roth B, Kribs A, Mehler K. Delivery room skin-to-skin contact in preterm infants affects long-term expression of stress response genes. Psychoneuroendocrinology. 2020 Dec;122:104883. doi: 10.1016/j.psyneuen.2020.104883. Epub 2020 Sep 24. PMID 33027708